CLINICAL TRIAL: NCT03448705
Title: A Phase I, Open-label to the Route of Administration, Single-blind to the ID Doses, Randomised, Active-controlled, Parallel Study to Evaluate the Safe Usability of 4Fluart ID Suspension for Injection in Adult Subjects
Brief Title: Safety of 4Fluart ID Suspension for Injection in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4Fluart-H-21
Record Dates: First submitted 2017-09-26; First posted 2018-02-28 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Human Influenza
Keywords: influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Injections

STUDY DESIGN:
Intervention Model Description: According to the objective, as well as the primary endpoints of the study, this is a Phase I study, open-label to the route of administration, single-blind to the ID doses, randomised, active-controlled that will be conducted in three parallel groups. Three visits will be performed in the study: on Day 0, Day 7-9 and Day 21-28. Pre-vaccination and post-vaccination serum samples are to be taken on Day 0 and Day 21-28. Adverse events will be documented between the enrollment and Day 21-28.
Who Masked: Participant
Masking Description: The study is single-blind (blinded for the participant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Study drug 1 (i.e. 4Fluart ID 1 µg/0.1 ml QIV) (Experimental): Vaccination of 12 subjects will be performed with the intradermal quadrivalent influenza vaccine containing 1 µg haemagglutinin per virus strain in 0.1 ml as a single dose.
  Interventions: Biological: 4Fluart ID suspension for injection study drug 1 µg/0.1 ml, influenza vaccine (whole virion, inactivated, adjuvanted)
- Group 2 - Study drug 2 (i.e. 4Fluart ID 2 µg/0.1 ml QIV) (Experimental): Vaccination of 12 subjects will be performed with the intradermal quadrivalent influenza vaccine containing 2 µg haemagglutinin per virus strain in 0.1 ml as a single dose.
  Interventions: Biological: 4Fluart ID suspension for injection study drug 2 µg/0.1 ml, influenza vaccine (whole virion, inactivated, adjuvanted)
- Group 3 - Comparator drug (i.e. 3Fluart IM 6 µg/0.5 ml TIV) (Active Comparator): Vaccination of 12 subjects will be performed with the intramuscular trivalent influenza vaccine containing 6 µg haemagglutinin per virus strain in 0.5 ml as a single dose.
  Interventions: Biological: 3Fluart suspension for injection, influenza vaccine (whole virion, inactivated, adjuvanted)

INTERVENTIONS:
Biological: 4Fluart ID suspension for injection study drug 1 µg/0.1 ml, influenza vaccine (whole virion, inactivated, adjuvanted) — Route of administration: intradermal, Dosage: 1 μg HA/strain / 0.1 ml, Package: 0.5 ml in one ampoule from which 0.1 ml is equal to a single dose, Dosage regimen: 1 x 0.1 ml, Treatment duration: single dose.
  Other Names: 4Fluart ID suspension for injection study drug; 4Fluart ID 1 µg/0.1 ml QIV
  Arms: Group 1 - Study drug 1 (i.e. 4Fluart ID 1 µg/0.1 ml QIV)
Biological: 4Fluart ID suspension for injection study drug 2 µg/0.1 ml, influenza vaccine (whole virion, inactivated, adjuvanted) — Route of administration: intradermal, Dosage: 2 μg HA/strain / 0.1 ml, Package: 0.5 ml in one ampoule from which 0.1 ml is equal to a single dose, Dosage regimen: 1 x 0.1 ml, Treatment duration: single dose.
  Other Names: 4Fluart ID suspension for injection study drug; 4Fluart ID 2 µg/0.1 ml QIV
  Arms: Group 2 - Study drug 2 (i.e. 4Fluart ID 2 µg/0.1 ml QIV)
Biological: 3Fluart suspension for injection, influenza vaccine (whole virion, inactivated, adjuvanted) — Route of administration: intramuscular, Dosage: 6 μg HA/strain / 0.5 ml, Package: 0.5 ml in one ampoule from which a total of 0.5 ml is equal to a single dose, Dosage regimen: 1 x 0.5 ml, Treatment duration: single dose.
  Other Names: 3Fluart suspension for injection; 3Fluart IM 6 µg/0.5 ml TIV
  Arms: Group 3 - Comparator drug (i.e. 3Fluart IM 6 µg/0.5 ml TIV)

SUMMARY:
The primary objective of the study is to evaluate the safe usability of the study drugs, i.e. 4Fluart ID 1 µg haemagglutinin (HA)/0.1 ml QIV and 4Fluart ID 2 µg haemagglutinin (HA)/0.1 ml QIV in terms of safety concerns emerged.

The secondary objective of the study is to further assess safety in terms of safety parameters, as well as to assess the immunogenicity of 4Fluart ID 1 µg haemagglutinin (HA)/0.1 ml QIV and 4Fluart ID 2 µg haemagglutinin (HA)/0.1 ml QIV in terms of immunogenicity parameters.

DETAILED DESCRIPTION:
Healthy volunteers (male and female) aged 18-59 years were enrolled into the study by signing subject information leaflet and informed consent form. After screening them, subjects complying with inclusion and exclusion criteria were included in the study, randomised and vaccinated with one of the investigational medicinal products assigned by the randomisation list.

Subjects were observed for thirty (30) minutes after vaccination for any immediate reactions. All adverse events (AEs) were collected from the enrolment to Day 21-28. Safety data between Day 0 and Day 7-9 were documented on a Diary card by each subject. Safety assessment were performed based on Day 7-9 and Day 21-28 safety data compared to the baseline on Day 0.

Blood samples for immunogenicity assays were collected immediately before vaccination on Day 0 (pre-vaccination blood samples) and on Day 21-28 (post-vaccination blood samples) in all subjects included in the study and complying with the study procedures. Immunogenicity were evaluated by hemagglutinin inhibition test in order to assess immune response 3-4 weeks after vaccination.

The assessment of safety and immunogenicity of 4Fluart ID 1 µg/0.1 ml QIV and 4Fluart ID 2 µg/0.1 ml QIV was performed in comparison to the authorised 3Fluart, i.e. 3Fluart intramuscular (IM) 6 µg/0.5 ml TIV.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons aged 18 to 59 years, determined on the day of enrolment from both sexes, mentally competent;
* Good health (as determined by vital signs and existing medical condition) or stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or insulin treated), the significance of which, in the opinion of the investigator, will not compromise the subject's participation in the study;
* Female volunteers of childbearing potential upon the decision of the investigator with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and to not become pregnant for the duration of the study;
* Capability of participants to understand and comply with planned study procedures;
* Participants provide written informed consent prior to initiation of study procedures;
* Absence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study. Pregnancy with regard to the total duration of the study.
* Hypersensitivity to the active substances or to any of the excipients, such as thiomersal, or any component that may be present in traces, such as egg (ovalbumin), formaldehyde, gentamicin, neomycin, vancomycin or ciprofloxacin determined prior to vaccination;
* Serious complications in the medical history with regard to any previous vaccination: encephalitis/encephalopathy, nonfebrile seizures, Guillain-Barré syndrome, vasculitis, neuritis, facial paresis determined prior to vaccination;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine determined prior to vaccination;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure with regard to the total duration of the study;
* Immunosuppressive therapy within 36 months prior to vaccination and with regard to the total duration of the study;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids with regard to the total duration of the study;
* Receipt of immunostimulants with regard to the total duration of the study;
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivate within 3 months prior to vaccination and with regard to the total duration of the study;
* Suspected or known HIV, Hepatitis-B virus (HBV) or Hepatitis-C virus (HCV) infection with regard to the total duration of the study;
* Acute disease and/or axillary temperature ≥37oC within 3 days prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination and with regard to the total duration of the study;
* Influenza vaccination (any kind) within 6 months prior to vaccination and with regard to the total duration of the study;
* Experimental drug therapy within 4 weeks prior to vaccination and with regard to the total duration of the study;
* Concomitant participation in another clinical study;
* Any condition which, may interfere with the evaluation of the study (including major protocol deviation with regard to the total duration of the study);
* Past or current psychiatric disease of the volunteer that upon judgement of the investigator may have an effect on the objective decision-making of the volunteer;
* Alcohol or drug abuse of the participant.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Safety in terms of safety concenrs emerged | Between 0 day (day of vaccination) and 21-28 days after vaccination
  Percentage of subjects reporting safety concerns following vaccination Measurement is based on the assessment of the study investigator by each subject

SECONDARY OUTCOMES:
Ratio of geometric mean anti-hemagglutinin antibody titres, for A/H1N1, A/H3N2, B strains | Between 0 day (day of vaccination) and 21-28 days after vaccination
  Ratio of Day 21-28 and Day 0 titres Anti-hemagglutinin antibodies are measured by hemagglutinin inhibition test
Percentage of subjects seroconverted based on anti-hemagglutinin antibody titres, for A/H1N1, A/H3N2, B strains | 0 days (day of vaccination) and 21-28 days after vaccination
  Seroconversion is defined as in subjects seronegative at baseline (i.e. HI titre <1:10 at Day 0) a post-vaccination HI titre ≥1:40, and in subjects seropositive at baseline (i.e. HI titre ≥1:10 at Day 0) as minimum of a 4-fold increase in post-vaccination HI titre Anti-hemagglutinin antibodies are measured by hemagglutinin inhibition test
Percentage of subjects seroprotected based on anti-hemagglutinin antibody titres, for A/H1N1, A/H3N2, B strains | 0 days (day of vaccination) and 21-28 days after vaccination
  The seroprotection rate is defined as a proportion of subjects with HI titre ≥1:40.
  Anti-hemagglutinin antibodies are measured by hemagglutinin inhibition test

CONTACTS AND LOCATIONS:
Overall Officials: Orsolya Gyurján, Study Director — Fluart Innovative Vaccines Ltd.
Locations (1):
- Drug Research Center, Balatonfüred, Veszprém megye, Hungary